CLINICAL TRIAL: NCT01250509
Title: Effects of Stress Reduction on Eating, Fat Distribution, and Cell Aging Among Overweight Women
Brief Title: Craving and Lifestyle Management Through Mindfulness Study
Acronym: CALMM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Mount Zion Health Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H11640-29259-03A; K01AT004199 (NIH)
Record Dates: First submitted 2010-11-23; First posted 2010-11-30 (Estimated); Results first posted 2013-02-18 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-01

CONDITIONS: Obesity
Keywords: Obesity; Mindfulness based stress reduction; Mindful eating; Stress; Overnutrition; Nutrition Disorders; Overweight; Body Weight; Signs and Symptoms
MeSH Terms: conditions — Obesity; Overnutrition; Nutrition Disorders; Overweight; Body Weight; Signs and Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CALMM (Experimental): Participants receiving the 'Craving and Lifestyle Management through Mindfulness' intervention, i.e. program that combines stress reduction with mindful eating practices.
  Interventions: Behavioral: Craving and Lifestyle Management through Mindfulness
- Waitlist Control (No Intervention): Participants were waitlisted for the intervention during the experimental phase.

INTERVENTIONS:
Behavioral: Craving and Lifestyle Management through Mindfulness — A preliminary, novel intervention was developed drawing on components from Mindfulness-Based Stress Reduction (MBSR), Mindfulness-Based Cognitive Therapy (MBCT), and Mindfulness-Based Eating Awareness Training (MB-EAT). The intervention program consisted of nine 2.5-hour classes and one 7-hour silent day of guided meditation practice after class 6.
  Arms: CALMM

SUMMARY:
The purpose of this study is to determine whether a mindfulness-based stress reduction and mindful eating program will lead to reductions in abdominal fat and total weight and improve cell aging in overweight and obese women compared to a waitlist control group.

DETAILED DESCRIPTION:
Obesity is the largest growing epidemic, with about 65% of Americans overweight (Flegal, Carroll et al. 2002). Obesity, in particular, abdominal obesity, confers increased risk for a host of diseases, including hypertension, Type 2 diabetes, and coronary heart disease, resulting in shortened life span (Fontaine, Redden et al. 2003). Psychological stress is widely cited anecdotally as a factor that causes people to engage in overeating, and studies provide strong evidence that stress can promote obesity. Stress induces selective preference of sweet, high-fat food and increases visceral fat depots. The telomere maintenance system (telomerase activity and telomere length)are markers of cellular aging and predict mortality (Cawthon et al, 2003)and have been linked to both psychological stress and components of the metabolic syndrome. The proposed study adapts a program called Mindfulness-Based Stress Reduction (MBSR) that has been shown to be effective in a variety of other stress-related conditions. Fifty overweight, pre-menopausal women at risk for the Metabolic Syndrome will be randomized in a 1:1 distribution to either a 3-month intervention to reduce stress and overeating [Craving and Lifestyle Management with Mindfulness (CALMM)] or wait list control group. The primary outcome measures include amounts of abdominal fat, weight, and telomerase activity. Data from this study are intended to provide pilot data for use in planning a larger randomized, controlled trial that will investigate the effects of the CALMM intervention on the metabolic and psychological processes assessed in this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal
* BMI (25 - 40)
* Weight < 300 lbs.
* Negative urine glucose test

Exclusion Criteria:

* Inability to provide informed consent
* Age < 21 or menopausal as determined by self-report
* DSM-IV diagnosis of an eating disorder
* Any substance abuse, mental health, or medical condition that, in the opinion of investigators, will make it difficult for the potential participant to participate in the intervention
* Factors that confound relations between stress and eating, including, drug abuse and use of medications containing corticosteroids.
* Diabetes
* Polycystic Ovary Syndrome
* CHD
* Breastfeeding (due to interference with stress hormone measurement)
* Non English speaker
* Pregnant as determined by pregnancy test at screening visit or planning to get pregnant in the next 6 months
* Previous MBSR training and/or current meditation, yoga, or other mind-body practice
* Initiation of new class of psychiatric medications in past 2 months.
* Currently on a weight loss diet

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2006-11; Primary Completion 2007-10 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Epel, PhD, Principal Investigator — UCSF Department of Psychiatry; Frederick Hecht, MD, Principal Investigator — UCSF Osher Center for Integrative Medicine; Jennifer Daubenmier, PhD, Principal Investigator — UCSF Osher Center for Integrative Medicine
Locations (1):
- UCSF Osher Center for Integrative Medicine, San Francisco, California, United States

REFERENCES:
- [Background] Baer RA, Smith GT, Allen KB. Assessment of mindfulness by self-report: the Kentucky inventory of mindfulness skills. Assessment. 2004 Sep;11(3):191-206. doi: 10.1177/1073191104268029. PMID 15358875
- [Background] Flegal KM, Carroll MD, Ogden CL, Johnson CL. Prevalence and trends in obesity among US adults, 1999-2000. JAMA. 2002 Oct 9;288(14):1723-7. doi: 10.1001/jama.288.14.1723. PMID 12365955
- [Background] Epel ES, McEwen B, Seeman T, Matthews K, Castellazzo G, Brownell KD, Bell J, Ickovics JR. Stress and body shape: stress-induced cortisol secretion is consistently greater among women with central fat. Psychosom Med. 2000 Sep-Oct;62(5):623-32. doi: 10.1097/00006842-200009000-00005. PMID 11020091
- [Background] Oliver G, Wardle J, Gibson EL. Stress and food choice: a laboratory study. Psychosom Med. 2000 Nov-Dec;62(6):853-65. doi: 10.1097/00006842-200011000-00016. PMID 11139006
- [Background] Boggiano MM, Chandler PC, Viana JB, Oswald KD, Maldonado CR, Wauford PK. Combined dieting and stress evoke exaggerated responses to opioids in binge-eating rats. Behav Neurosci. 2005 Oct;119(5):1207-14. doi: 10.1037/0735-7044.119.5.1207. PMID 16300427
- [Background] Yusuf S, Hawken S, Ounpuu S, Bautista L, Franzosi MG, Commerford P, Lang CC, Rumboldt Z, Onen CL, Lisheng L, Tanomsup S, Wangai P Jr, Razak F, Sharma AM, Anand SS; INTERHEART Study Investigators. Obesity and the risk of myocardial infarction in 27,000 participants from 52 countries: a case-control study. Lancet. 2005 Nov 5;366(9497):1640-9. doi: 10.1016/S0140-6736(05)67663-5. PMID 16271645
- [Background] Epel E, Lapidus R, McEwen B, Brownell K. Stress may add bite to appetite in women: a laboratory study of stress-induced cortisol and eating behavior. Psychoneuroendocrinology. 2001 Jan;26(1):37-49. doi: 10.1016/s0306-4530(00)00035-4. PMID 11070333
- [Background] Epel E, Jimenez S, Brownell K, Stroud L, Stoney C, Niaura R. Are stress eaters at risk for the metabolic syndrome? Ann N Y Acad Sci. 2004 Dec;1032:208-10. doi: 10.1196/annals.1314.022. PMID 15677412
- [Background] Rebuffe-Scrive M, Walsh UA, McEwen B, Rodin J. Effect of chronic stress and exogenous glucocorticoids on regional fat distribution and metabolism. Physiol Behav. 1992 Sep;52(3):583-90. doi: 10.1016/0031-9384(92)90351-2. PMID 1409924
- [Background] Rosmond R. Role of stress in the pathogenesis of the metabolic syndrome. Psychoneuroendocrinology. 2005 Jan;30(1):1-10. doi: 10.1016/j.psyneuen.2004.05.007. PMID 15358437
- [Background] Roemmich JN, Wright SM, Epstein LH. Dietary restraint and stress-induced snacking in youth. Obes Res. 2002 Nov;10(11):1120-6. doi: 10.1038/oby.2002.152. PMID 12429875

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Female participants were recruited through media outlets and flyers posted in the San Francisco Bay Area. Three hundred twenty-two potential participants were screened for eligibility from November 2006 to March 2007.
Pre-assignment Details: Fifty-three met eligibility criteria and chose to enroll, and 47 went on to the randomization stage. Before randomization, 5 participants dropped due to time constaints and 1 dropped due to illness.
Groups:
- CALMM: Participants receiving CALMM intervention, i.e. program that combines stress reduction with mindful eating practices.
Period: Overall Study
Arm/Group | CALMM | Waitlist Control
Started | 24 | 23
Completed | 19 | 21
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CALMM | Waitlist Control | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 23 | 47
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 40.4 (8.0) | 41.4 (6.7) | 40.9 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 47
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 23 | 47

OUTCOME MEASURES:

1. Primary Outcome: Change in Abdominal Fat
Description: Whole-body dual energy X-ray absorptiometry (DEXA) scans were performed to assess body fat distribution. The DEXA densitometry (GE Healthcare Lunar Prodigy, Madison, Wis, USA) was adjusted to the fan beam mode and EnCore software version 9.15 was used. The primary region of interest was fat tissue from a rectangular region in the abdominal area defined by the upper boundary of the second lumbar vertebra to the lower edge of the fourth lumbar vertebra. The vertical sides were defined as the continuation of the lateral sides of the rib cage.
Time Frame: Change from Baseline in Abdominal Fat (baseline and 4 months)
Population: Intent-to-treat analyses were conducted. Assuming participants lost to followup did not change over time, missing data at postintervention were imputed using preintervention values.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | CALMM | Waitlist
Number analyzed (Participants) | 24 | 23
grams | 68.2 (318.9) | 50.0 (305.4)

2. Secondary Outcome: Weight
Time Frame: Change in Weight (baseline and 4 months)
Population: Intention to treat analysis was conducted. Assuming participants lost to followup did not change over time, missing data at postintervention were imputed using preintervention values.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | CALMM | Waitlist Control
Number analyzed (Participants) | 24 | 23
kg | -0.03 (2.7) | 0.38 (1.9)

3. Secondary Outcome: Telomerase Activity
Description: Cryopreserved peripheral blood nuclear cells (PBMCs) were thawed and live cells counted using a hemocytometer by the Trypan blue exclusion method. For each sample, an extract of 5000 cells per microliter was made and two concentrations, corresponding to 5000 and 10,000 cells, were assayed for each sample to ensure the assay was in the linear range. Telomerase activity was assayed by the Telomerase Repeat Amplification Protocol (TRAP) using a commercial kit (TRAPeze, Telomerase Detection kit, Upstate/ CHEMICON, Temecula, CA). Baseline and post-intervention samples for the same participant were assayed in the same batch and run on the same gel to eliminate any differences caused by reaction or procedural batch-to-batch variations. Technicians were blind to group assignment. Telomerase activity is defined as 1 unit = the amount of product from one 293T cell/10,000 PBMCs, and was quantified using the software ImageQuant 5.2 (GE Healthcare, Piscataway, NJ).
Time Frame: Change from Baseline in Telomerase Activity at 4 months
Population: Intention-to-treat analysis was conducted.
Measure: Mean (Standard Deviation); unit: Standard arbitrary units, see above
Arm/Group | CALMM | Waitlist Control
Number analyzed (Participants) | 19 | 18
Standard arbitrary units, see above | 0.24 (0.5) | 0.15 (0.3)

4. Secondary Outcome: Change in Psychological Stress (Baseline and 4 Months)
Description: The 10-item Perceived Stress Scale was used to evaluate perception of stressful events over the past month by using a 5-point Likert scale (0 = never to 4 = very often) (Cohen et al., 1983). The mean of the ten items was used in analysis. Higher scores indicate greater perceived stress.
Time Frame: Change from Baseline in Psychological Stress
Population: An intention-to-treat analysis was conducted. Assuming participants lost to followup did not change over time, missing data at postintervention were imputed using preintervention values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CALMM | Waitlist Control
Number analyzed (Participants) | 24 | 23
units on a scale | -0.20 (0.5) | 0.03 (0.6)

ADVERSE EVENTS:
Arm/Group | CALMM | Waitlist Control
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 0/47 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes